CLINICAL TRIAL: NCT05513976
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of SHR4640 Tablets Combined With Febuxostat Tablets in the Treatment of Primary Gout and Hyperuricemia Subjects With Inadequate Control on Febuxostat
Brief Title: Clinical Study of SHR4640 Tablets Combined With Febuxostat Tablets in the Treatment of Primary Gout and Hyperuricemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR4640-203
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Primary Gout and Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — ruzinurad; Febuxostat

STUDY DESIGN:
Intervention Model Description: SHR4640 VS. Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- treatment group A (Experimental)
  Interventions: Drug: SHR4640 tablet; Drug: febuxostat tablet
- treatment group B (Experimental)
  Interventions: Drug: SHR4640 tablet; Drug: febuxostat tablet
- treatment group C (Placebo Comparator)
  Interventions: Drug: febuxostat tablet; Drug: SHR4640 placebo tablet

INTERVENTIONS:
Drug: SHR4640 tablet — SHR4640 tablet 5mg
  Arms: treatment group A
Drug: SHR4640 tablet — SHR4640 tablet 10mg
  Arms: treatment group B
Drug: febuxostat tablet — febuxostat tablet 40mg or 60mg or 80mg based on prior medication
Drug: SHR4640 placebo tablet — SHR4640 placebo tablet 5 or 10mg
  Arms: treatment group C

SUMMARY:
SHR4640 tablets is a highly selective and potent URAT1 inhibitors,study number is SHR4640-203. The primary purpose of the study is to evaluate the efficacy and safety of the combination of SHR4640 and febuxostat compared with placebo and febuxostat in primary gout and hyperuricemia subjects with inadequate control on febuxostat for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent, understood the procedures and methods of the study, and was willing to complete the study strictly in accordance with the clinical trial protocol;
2. The screening age should be 18-65 years old (including both ends), male or female; 3. Receiving febuxostat dose ≥40mg/ day, not more than 80mg/ day, stable dose for ≥6 weeks, fasting serum uric acid ≥390µmol/L at screening; 4. Meet the 1977 or 2015 American College of Rheumatology (ACR) criteria for classification of gout; 5、18kg/m2≤ Body weight Mass index (BMI) ≤35kg/m2.

Exclusion Criteria:

1. General Situation:

   * 1) Pregnant or lactating women;
   * 2) Refusal or use of medically unapproved contraceptive measures by fertile women or men (except for non-fertile partners) within 3 months of screening to the last medication for men and 6 months for women;
   * 3) The average daily alcohol intake in the 1 month prior to screening was more than 14g (e.g., 145mL wine, 497mL beer, or 43mL low-alcohol liquor) for women and more than 28g (e.g., 290mL wine, 994mL beer, or 86mL low-alcohol liquor) for men;
   * 4) Drug abusers;
   * 5) Subjects whose compliance is considered by the investigator to be poor and affect the evaluation of the safety and efficacy of the trial drug.
2. The following conditions occurred in the laboratory examination within 3 weeks before randomization:

   * 1) upper limit of alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) and/or total bilirubin (T-Bil);
   * 2) Serum creatinine was calculated using simplified Diet adjustment for Kidney Disease (MDRD) formula and eGFR was less than 45mL/ (min×1.73m2).
   * 3) Glycosylated hemoglobin (HbA1c) ≥8%;
   * 4) Having active hepatitis B [hepatitis B surface antigen (HBsAg) positive and HBV deoxyribonucleic acid (HBV-DNA) ≥500 IU/mL or 2500 copies/mL], or anti-hepatitis C virus (HCV) antibody positive, or human immunodeficiency virus (HIV) antibody positive, Or a positive syphilis antibody test;
   * 5) White blood cell < 3.0×109/L, and/or hemoglobin < 90 g/L, and/or platelet < 80×109/L.
3. Any of the following medical history or comorbidities:

   * 1) Allergy, allergy to SHR4640 or any component of SHR4640, or previous intolerance to febuxostat or contraindications;
   * 2) Secondary hyperuricemia caused by tumors, chronic kidney diseases, blood diseases, drugs and other reasons;
   * 3) There are other joint lesions that researchers believe may confuse gouty arthritis, such as rheumatoid arthritis, pyogenic arthritis, traumatic arthritis, psoriatic arthritis, pseudogout, systemic lupus erythematosus, or joint lesions caused by chemotherapy, radiotherapy, chronic lead poisoning, acute obstructive nephropathy, etc.
   * 4) Urinary calculi were detected or suspected by B-ultrasound within 3 weeks before randomization;
   * 5) Gout attack within 2 weeks before randomization;
   * 6) History of active peptic ulcer within 1 year before screening or active peptic ulcer at screening;
   * 7) History of xanthine urine;
   * 8) The presence of malignancy, or a history of malignancy within 5 years prior to screening (except for treated non-melanoma of the skin without signs of recurrence, and resected cervical intraepithelial neoplasia);
   * 9) History of chronic infection or recurrent infection within 1 year before screening; Or a serious infection (including but not limited to hepatitis, sepsis, pneumonia, pyelonephritis, etc.) or infection leading to hospitalization in the 3 months prior to screening; Or an infection that was treated with intravenous antibiotics before screening; Or open draining wounds or ulcers at the time of screening;
   * 10) Patients who need to use immunosuppressive agents for systemic therapy;
   * 11) Moderate to severe congestive heart failure (New York Heart Association class III or IV);
   * 12) Myocardial infarction, unstable angina pectoris, percutaneous transluminal coronary angioplasty, coronary artery bypass grafting, brain infarction, cerebral hemorrhage, subarachnoid hemorrhage, or transient ischemic attack, and other cardiovascular and cerebrovascular events leading to hospitalization occurred within 1 year before screening;
   * 13) Poorly controlled hypertension [systolic blood pressure (SBP) ≥180mmHg and/or diastolic blood pressure (DBP) ≥110mmHg at rest, reconfirmed];
   * 14) combined with other serious or poorly controlled diseases;
   * 15) Patients who had undergone major surgery within 3 months prior to surgery, or had not recovered from surgery, or planned to undergo major surgery during the study period;
   * 16) Blood donation (or blood loss) and blood donation (or blood loss) ≥400 mL within 3 months before screening, or receiving blood transfusion.
4. Use any of the following drugs or participate in clinical trials:

   * 1) Participated in any investigational drug (including investigational vaccine) clinical trial and used investigational drug within 3 months before screening or within the half-life of 5 investigational drugs (whichever is longer);
   * 2) Participated in any clinical trial of medical device within 3 months prior to screening (excluding failed screening subjects);
   * 3) Use other uric acid lowering drugs (allopurinol, benzbromarone, and recombinant uricase) within 6 weeks before screening;
   * 4) Drugs that interact with febuxostat (theophylline, azathioprine, mercaptopurine) were used within 6 weeks before screening;
   * 5) Within 6 weeks before screening, the daily dose of aspirin was more than 100mg or the dose was unstable;
   * 6) Use any diuretic within 2 weeks before randomization;
   * 7) Blood pressure, lipid-lowering and glucose-lowering drugs with unstable dose were used within 2 weeks before randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with serum uric acid ≤360μmol/L | After 12 weeks of treatment

SECONDARY OUTCOMES:
Proportion of subjects with serum uric acid ≤ 300μmol/L (response) | After 12 weeks of treatment
Proportion of subjects with serum uric acid ≤360μmol/L at the last two tests at 12 weeks of double-blind treatment | After 12 weeks of treatment
Percentage change in serum uric acid from baseline at each visit | within 12 weeks of double-blind treatment
Changes in serum uric acid from baseline at each visit | within 12 weeks of double-blind treatment
Proportion of subjects with serum uric acid ≤360μmol/L at each visit | within 12 weeks of double-blind treatment

IPD SHARING:
Plan to Share IPD: Undecided